CLINICAL TRIAL: NCT02859831
Title: Fungal Contamination of a Hospital Water System With Fusarium App.: Prospective Environmental and Medical Surveillance During a Construction Period
Brief Title: Sautour PHRC IR 2008
Acronym: SautourPHRCI08
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Sautour PHRC IR 2008
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Mycosis
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- with construction work
  Interventions: Other: water samples
- without construction work
  Interventions: Other: water samples

INTERVENTIONS:
Other: water samples

SUMMARY:
Fusarium are microscopic filamentous fungi that live as saprobiontics in outside environments. They are found in the soil, the air, in water and on numerous plants. The frequency of fusariosis is currently increasing and Fusarium-related mycoses are the 3rd most frequent invasive mycoses. Most cases have been reported in the United States, in France, in Italy and in Brazil. A few epidemiological studies have shown the role of water in the appearance of mycoses in highly immunodepressed patients. Few studies have focused on the role of water in the transmission of mycoses in hospitals. The aim of this prospective study is to describe, in time and pace, the contamination by Fusarium sp. in the water of two different hospitals (Dijon, Nancy), by taking into account factors such as seasons and major works (reconstruction of a hospital). In each hospital, one reconstruction site will be compared with a site not under reconstruction (control).

Water samples will be taken from the rooms of hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

all patients with new-onset fusariosis in the Adult Haematology, Internal Medicinie, Digestive Surgery and Rheumatology Departments

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: water samples from the rooms of hospitalized patients in 4 departments of Dijon and Nancy CHU
Sampling Method: Non-Probability Sample
Enrollment: 551 (Actual)
Dates: Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Presence of Fusarium sp | every week throughout the study, thus over 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France